CLINICAL TRIAL: NCT03558438
Title: Spanish Cohort of Patients with HIV Infection Older Than 50 Years for the Study of Fragility and Physical Function
Acronym: FUNCFRAIL
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Other Study IDs: GESIDA 9817
Record Dates: First submitted 2018-05-25; First posted 2018-06-15 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections; Frail Older Adults
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Markers of mitochondrial function, of naive cells, memory and recent immigrants of the thymus, of immunoactivation, immunosenescence, activation / exhaustion and proliferation and Telomere measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV patients older than 50 years: Spanish cohort of patients with HIV infection older tha 50 years old.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
It's a prospective observational study to assess frailty and physical function

DETAILED DESCRIPTION:
We stimate to recruit 1120 patients older tan 50 years to assess frailty and define a simplified fragility index

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed HIV + infection.
2. Patients aged ≥ 50 years at the time of starting the study, followed in the Infectious-HIV consultations of the centers participants.

   This limit has been chosen because it is accepted by the scientific community for define the elderly patient in patients with HIV infection.
3. Have signed the informed consent and be willing to comply with the study visits.

Exclusion Criteria:

1. Have an established disability that does not allow you to walk.
2. Patients who can not comply with the visits and study procedures or who are not usually followed at the center.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV infection older ythan 50 year sold who are followed in the consultations of the center participants
Sampling Method: Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To know the prevalence of frailty in the population over 50 years old with HIV infection according to Fried's fragility phenotype | Change from basal to year 5
  Fragility is defined according to the 5 Fried criteria:
  * Involuntary weight loss: (> 4.5Kg in the last year)
  * Declined mood: through two questions from the Scale for Depression of the Center for Epidemiological Studies (CES-D).
  * Speed of walking adjusted for height and sex,
  * Weekly physical activity adjusted by sex.
  * Muscle weakness according to manual grip strength adjusted for BMI and sex.
Define a new simplified fragility index for the elderly patients with HIV infection easily applicable in clinical routine practice | Year 5
  The simplified fragility index for the elderly patient with HIV infection can not be defined a priori, so a multivariate logistic regression analysis will be performed for those variables that are associated with fragility in the analysis univariate, which will allow us to determine the variables that are associated in a independent with fragility, which will be with which we will define the fragility index simplified. Fragility will be treated as a binary variable: pre-fragile and robust will form a group that will serve as control. The fragility phenotype defined by the 5 Fried criteria will be considered the gold standard test to measure fragility when validating the simplified fragility screening test specific for elderly patients with HIV infection that we want to define
To study the prognostic value of the CD4 / CD8 ratio in relation to frailty | Change from Basal to Year 5
Analyze the relationship between exposure time to different families of antiretroviral drugs with fragility. | Change from Basal to Year 5
Define fragility biomarkers | Change from Basal to Year 5
  immunological profile, oxidative damage, microbiome.

SECONDARY OUTCOMES:
Know the functional situation and the risk of functional deterioration of the population over 50 years of age with HIV infection in our cohort | Year 1, year 2, year 3, year 4 and year 5
Analyze the possible association of fragility in this population group with the comorbidity and the presence of other geriatric syndromes | Year 1, year 2, year 3, year 4 and year 5
To know the prevalence of other geriatric syndromes | Year 1, year 2, year 3, year 4 and year 5
  polypharmacy, falls, cognitive impairment, depression, risk of malnutrition.
To know the risk of fragility fractures in the population over 50 years old with HIV infection in our cohort | Year 1, year 2, year 3, year 4 and year 5
To analyze the possible association of bone fragility with the presence of the syndrome clinical of fragility in this population group | Year 1, year 2, year 3, year 4 and year 5

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - Hospital Reina Sofia, Córdoba, Córdoba
  - Hospital de Donostia, Donostia / San Sebastian, Donostia
  - Clínico San Carlos, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Univ. La Paz, Madrid, Madrid
  - Hospital de Santiago, Santiago de Compostela, Santiago de Compostela
  - Hospital Clínic de Valencia, Valencia, Valencia
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital de Guadalajara, Guadalajara
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Puerta de Hierro, Madrid

REFERENCES:
- [Derived] Branas F, Torralba M, Antela A, Vergas J, Ramirez M, Ryan P, Dronda F, Galindo MJ, Machuca I, Bustinduy MJ, Cabello A, Montes ML, Sanchez-Conde M; FUNCFRAIL study group. Effects of frailty, geriatric syndromes, and comorbidity on mortality and quality of life in older adults with HIV. BMC Geriatr. 2023 Jan 3;23(1):4. doi: 10.1186/s12877-022-03719-8. PMID 36597036